CLINICAL TRIAL: NCT02912780
Title: Introduction of Microsystems in a Level 3 Neonatal Intensive Care Unit - an Interprofessional Approach
Brief Title: Introduction of Microsystems in a Level 3 Neonatal Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Christoph Fusch, Professor, McMaster Children's Hospital
Other Study IDs: COHORT2013
Record Dates: First submitted 2016-09-14; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Stress, Psychological; Inflammatory Bowel Diseases; Lung Diseases; Infant Nutrition Disorders; Eye Manifestations; Neurodevelopmental Disorders
MeSH Terms: conditions — Stress, Psychological; Inflammatory Bowel Diseases; Lung Diseases; Infant Nutrition Disorders; Eye Manifestations; Neurodevelopmental Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The advancement in life-saving technologies and clinical expertise in the care of extremely premature infants, have resulted in the development of large neonatal intensive care units (NICU). It has been suggested that reconstruction of megaunits of neonatal intensive care to smaller care units with specific patient population and clinical team providers will be essential to maintain optimal teamwork, quality of care and patient outcome.

Despite the growing knowledge around the need for reconstruction of large NICUs to smaller units of care, there is no evidence regarding the safety and efficacy of microsystem model of care on the key aspects of health care. At the McMaster Children's Hospital (MCH), we planned a change from standard model of care to the microsystem model of care and therefore we aimed to prospectively assess the effect of this organizational change on the variable aspects of health care.

A working group met weekly to formulate the implementation planning, to review the adaptation and adjustment process and to ascertain the quality of implementation following the initiation of the microsystem model.

The study was retrospectively registered.

ELIGIBILITY:
Inclusion criteria:

* All preterm and term infants admitted to McMaster Children's Hospital NICU

Exclusion criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm and term infants
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of stress level of Health Care Professional - Salivary cortisol (ng/dL) | once every week, up to 3 month corrected age
Change of stress level of Parents - Salivary cortisol (ng/dL) | once every week, up to 3 month corrected age
Change of stress level of Patients - Salivary cortisol (ng/dL) | once every week, up to 3 month corrected age
Length of stay - days | up to 3 month corrected age
Incidence of necrotizing enterocolitis | up to 3 month corrected age
Incidence of retinopathia of prematurity | up to 3 month corrected age
Incidence of bronchopulmonary dysplasia | up to 3 month corrected age
Incidence of sepsis | up to 3 month corrected age
Duration of mechanical ventilation - days | up to 3 month corrected age
Time of feed initiation - days | up to 3 month corrected age
Time to full feed - days | up to 3 month corrected age
Number of days with parenteral nutrition | up to 3 month corrected age
Bayley scale - Psychomotor Developmental Index | up to 3 month corrected age
Bayley scale - Mental Developmental Index | up to 3 month corrected age
Number of changes in the primary health care professionals | up to 3 month corrected age
Noise level (decibel) | up to 3 month corrected age
use of resources (lab tests, X-rays, microbiological tests) | up to 3 month corrected age
  number of procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Science, McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Helou S, Samiee-Zafarghandy S, Fusch G, Wahab MG, Aliberti L, Bakry A, Barnard D, Doucette J, El Gouhary E, Marrin M, Meyer CL, Mukerji A, Nwebube A, Pogorzelski D, Pugh E, Schattauer K, Shah J, Shivananda S, Thomas S, Twiss J, Williams C, Dutta S, Fusch C. Introduction of microsystems in a level 3 neonatal intensive care unit-an interprofessional approach. BMC Health Serv Res. 2017 Jan 21;17(1):61. doi: 10.1186/s12913-017-1989-6. PMID 28109276